CLINICAL TRIAL: NCT05802199
Title: Quantitative Detection Efficiency of Ultrasound Derived Fat Fraction (UDFF) as a Non-invasive Alternative for Nonalcoholic Fatty Liver Disease (CHESS2303): a Multicenter Prospective Study
Brief Title: Quantitative Detection Efficiency of UDFF for Nonalcoholic Fatty Liver Disease
Acronym: UDFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Zhongda Hospital (Other); Zhejiang University (Other); Lishui Country People's Hospital (Other); Shandong Public Health Clinical Center (Other Government); Affiliated Hangzhou Xixi Hospital, Zhejiang University School of Medicine (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Second Hospital of Anhui Medical University (Other); The People's Hospital of Bozhou (Unknown); The First Affiliated Hospital of Xiamen University (Other); The First Hospital of Jilin University (Other); Kliniken Hirslanden Beau Site, Salem und Permancence (Unknown); Third People's Hospital of Zhenjiang, Jiangsu University (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHESS2303
Record Dates: First submitted 2023-03-14; First posted 2023-04-06 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease (NAFLD); ultrasound-derived fat fraction (UDFF); hepatic fibrosis; point shear wave elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Patients were fulfilled diagnosis of non-alcoholic fatty liver disease based on radiological and clinical manifestation.
  Patients were fulfilled diagnosis of hepatic fibrosis based on radiological and clinical manifestation.
  Interventions: Diagnostic Test: Hepatic fat fraction and hepatic fibrosis
- Validation cohort: Patients were fulfilled diagnosis of non-alcoholic fatty liver disease based on radiological and clinical manifestation.
  Patients were fulfilled diagnosis of hepatic fibrosis based on radiological and clinical manifestation.
  Interventions: Diagnostic Test: Hepatic fat fraction and hepatic fibrosis

INTERVENTIONS:
Diagnostic Test: Hepatic fat fraction and hepatic fibrosis — All patients underwent measurement of UDFF for hepatic fat fraction and auto-pSWE for hepatic fibrosis.
  All patients underwent measurement of MRI-PDFF for hepatic fat fraction and MRE for hepatic fibrosis as reference standard.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease worldwide, affecting more than 25 % of the population globally. Approximately 20 % - 25 % of NAFLD patients can develop nonalcoholic steatohepatitis (NASH), which leads to more rapid progression from fibrosis to cirrhosis, and even liver failure or hepatocellular carcinoma (HCC). Early detection and treatment may halt or reverse NAFLD progression.

Although liver biopsy has been the well-accepted clinical reference standard for both diagnosis and staging of the different histological changes in NAFLD, this procedure is invasive with complications such as bleeding and infection, and is unreliable for quantifying steatosis due to sampling errors. Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) currently has been accepted as the preferred alternative to the histological assessment of hepatic steatosis in patients with NAFLD. Magnetic resonance elastography (MRE) provide additional information of inflammation and fibrotic components of NAFLD. However, important limitations hinder the widespread clinical application of MRI, including high cost, low availability, long scan times and exclusion of patients with metal implants.

Ultrasound (US) has been recommended by several guidelines as the first-line screening tool for patients at risk of NAFLD. The developed ultrasound-derived fat fraction (UDFF) is designed to assess hepatic steatosis by estimating the frequency-dependent attenuation coefficient (AC) and backscatter coefficient (BSC) through processing acoustic radiofrequency (RF) signals returned from the liver tissue as fat vesicles in hepatocytes have a different characteristic impedance compared to normal liver tissue. UDFF is available on the Acuson Sequoia ultrasound system (Simens Healthineers, Mountain View, CA, USA), with reference to integrated phantom data to correct for system impact, and produces a UDFF value presented as a fat fraction (%), which is potentially related to MRI-PDFF and can be directly compared with MRI-PDFF. In addition, automatic point shear wave elastography (auto-pSWE) is available on the Acuson Sequoia ultrasound system to obtain liver stiffness measurement (LSM) for assessing hepatic fibrosis, simultaneously with UDFF measurement. The prospective, multicenter study aims to evaluate the efficiency of UDFF as a quantitative non-invasive alternative for NAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease worldwide characterized by excessive accumulation of triglycerides in hepatocytes and subsequent steatosis, affecting more than 25 % of the population globally. Approximately 20 % - 25 % of NAFLD patients can develop nonalcoholic steatohepatitis (NASH), which leads to more rapid progression from fibrosis to cirrhosis, and even liver failure or hepatocellular carcinoma (HCC). NALFD is strongly associated with metabolic risk factors, such as obesity, cardiovascular disease, and diabetes mellitus. Early detection and treatment may halt or reverse NAFLD progression. However, the occurrence and progression of steatosis and fibrosis had no obvious clinical symptoms, resulting in a difficulty of early diagnose and grade individuals with NAFLD clinically.

Although liver biopsy has been the well-accepted clinical reference standard for both diagnosis and staging of the different histological changes in NAFLD, this procedure is invasive with complications such as bleeding and infection, and is unreliable for quantifying steatosis due to sampling errors. Several imaging modalities have been used to diagnose and grade hepatic steatosis. Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) currently has been accepted as the preferred alternative to the histological assessment of hepatic steatosis in patients with NAFLD. Magnetic resonance elastography (MRE) provide additional information of inflammation and fibrotic components of NAFLD. However, important limitations hinder the widespread clinical application of MRI, including high cost, low availability, long scan times and exclusion of patients with metal implants.

Ultrasound (US) has been recommended by several guidelines as the first-line screening tool for patients at risk of NAFLD. The most commonly used noninvasive method that quantifies the amount of fat in the liver is the controlled attenuation parameter, and more than 10% of steatosis can be distinguished. The disadvantages of this technique are that the liver morphological changes cannot be assessed simultaneously and poor performance in patients with higher body mass indices, leading to a failure rate of measurement ranged of 7.7 % - 14.0 %.

The developed ultrasound-derived fat fraction (UDFF) is designed to assess hepatic steatosis by estimating the frequency-dependent attenuation coefficient (AC) and backscatter coefficient (BSC) through processing acoustic radiofrequency (RF) signals returned from the liver tissue as fat vesicles in hepatocytes have a different characteristic impedance compared to normal liver tissue. UDFF is available on the Acuson Sequoia ultrasound system (Simens Healthineers, Mountain View, CA, USA), with reference to integrated phantom data to correct for system impact, and produces a UDFF value presented as a fat fraction (%), which is potentially related to MRI-PDFF and can be directly compared with MRI-PDFF. In addition, automatic point shear wave elastography (auto-pSWE) is available on the Acuson Sequoia ultrasound system to obtain liver stiffness measurement (LSM) for assessing hepatic fibrosis, simultaneously with UDFF measurement. The prospective, multicenter study aims to evaluate the efficiency of UDFF as a quantitative non-invasive alternative for NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age.
2. fulfilled diagnosis of non-alcoholic fatty liver disease based on radiological (MRI-PDFF values > 5%) and clinical manifestation.
3. fulfilled diagnosis of hepatic fibrosis with non-alcoholic fatty liver disease based on radiological (LSM by MRE > 3.02kPa) and clinical manifestation.
4. Willing to participate in this research and sign the informed consent.

Exclusion Criteria:

1. with liver dysfunction at the terminal stage or are ready for liver transplantation.
2. with viral hepatitis, autoimmune hepatitis, and alpha-1-antitrypsin deficiency.
3. history of excessive drinking (the amount of alcohol consumed by women is more than 140 grams per week, and that of men is more than 210 grams per week).
4. unable to cooperate with ultrasound examinations.
5. have taken liver damage drugs within the past six months.
6. with massive ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were fulfilled diagnosis of non-alcoholic fatty liver disease based on radiological and clinical manifestation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficiency of UDFF (in %) for hepatic steatosis in comparison with MRI-PDFF (in %). | 1 years
  Evaluate the diagnosis performance of ultrasound-derived fat fraction (UDFF) as a quantitative non-invasive alternative for diagnosing and grading of hepatic steatosis in NAFLD patients, taking MRI-PDFF as the reference standard.

SECONDARY OUTCOMES:
The efficiency of auto-pSWE (in kPa) for hepatic fibrosis in comparison with MRE (in kPa). | 1 years
  Evaluate the diagnosis performance of auto-pSWE as a quantitative non-invasive alternative for diagnosing and grading of hepatic fibrosis in NAFLD patients, taking MRE as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangao Fan, M.D., Study Chair — Xinhua Hospital, Shanghai Jiaotong University School of Medicine; Xiaolong Qi, M.D., Principal Investigator — Zhongda Hospital; Yi Dong, M.D., Study Director — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (14):
- China (13):
  - The People's Hospital of Bozhou, Bozhou, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhe Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Affiliated Hangzhou Xixi Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Kliniken Hirslanden Beau Site, Salem und Permancence, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ferraioli G, Berzigotti A, Barr RG, Choi BI, Cui XW, Dong Y, Gilja OH, Lee JY, Lee DH, Moriyasu F, Piscaglia F, Sugimoto K, Wong GL, Wong VW, Dietrich CF. Quantification of Liver Fat Content with Ultrasound: A WFUMB Position Paper. Ultrasound Med Biol. 2021 Oct;47(10):2803-2820. doi: 10.1016/j.ultrasmedbio.2021.06.002. Epub 2021 Jul 18. PMID 34284932
- [Result] Sanyal AJ, Brunt EM, Kleiner DE, Kowdley KV, Chalasani N, Lavine JE, Ratziu V, McCullough A. Endpoints and clinical trial design for nonalcoholic steatohepatitis. Hepatology. 2011 Jul;54(1):344-53. doi: 10.1002/hep.24376. PMID 21520200
- [Result] Simon TG, Roelstraete B, Khalili H, Hagstrom H, Ludvigsson JF. Mortality in biopsy-confirmed nonalcoholic fatty liver disease: results from a nationwide cohort. Gut. 2021 Jul;70(7):1375-1382. doi: 10.1136/gutjnl-2020-322786. Epub 2020 Oct 9. PMID 33037056
- [Result] Zhang MH, Li J, Zhu XY, Zhang YQ, Ye ST, Leng YR, Yang T, Zhang H, Kong LY. Physalin B ameliorates nonalcoholic steatohepatitis by stimulating autophagy and NRF2 activation mediated improvement in oxidative stress. Free Radic Biol Med. 2021 Feb 20;164:1-12. doi: 10.1016/j.freeradbiomed.2020.12.020. Epub 2021 Jan 1. PMID 33388433
- [Result] Chitturi S, Farrell GC, Hashimoto E, Saibara T, Lau GK, Sollano JD; Asia-Pacific Working Party on NAFLD. Non-alcoholic fatty liver disease in the Asia-Pacific region: definitions and overview of proposed guidelines. J Gastroenterol Hepatol. 2007 Jun;22(6):778-87. doi: 10.1111/j.1440-1746.2007.05001.x. PMID 17565630
- [Result] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. Diabetologia. 2016 Jun;59(6):1121-40. doi: 10.1007/s00125-016-3902-y. No abstract available. PMID 27053230
- [Result] Kim SH, Lee JM, Kim JH, Kim KG, Han JK, Lee KH, Park SH, Yi NJ, Suh KS, An SK, Kim YJ, Son KR, Lee HS, Choi BI. Appropriateness of a donor liver with respect to macrosteatosis: application of artificial neural networks to US images--initial experience. Radiology. 2005 Mar;234(3):793-803. doi: 10.1148/radiol.2343040142. Epub 2005 Jan 21. PMID 15665225
- [Result] Hernaez R, Lazo M, Bonekamp S, Kamel I, Brancati FL, Guallar E, Clark JM. Diagnostic accuracy and reliability of ultrasonography for the detection of fatty liver: a meta-analysis. Hepatology. 2011 Sep 2;54(3):1082-1090. doi: 10.1002/hep.24452. PMID 21618575
- [Result] Dasarathy S, Dasarathy J, Khiyami A, Joseph R, Lopez R, McCullough AJ. Validity of real time ultrasound in the diagnosis of hepatic steatosis: a prospective study. J Hepatol. 2009 Dec;51(6):1061-7. doi: 10.1016/j.jhep.2009.09.001. Epub 2009 Sep 20. PMID 19846234
- [Result] Marshall RH, Eissa M, Bluth EI, Gulotta PM, Davis NK. Hepatorenal index as an accurate, simple, and effective tool in screening for steatosis. AJR Am J Roentgenol. 2012 Nov;199(5):997-1002. doi: 10.2214/AJR.11.6677. PMID 23096171
- [Result] Webb M, Yeshua H, Zelber-Sagi S, Santo E, Brazowski E, Halpern Z, Oren R. Diagnostic value of a computerized hepatorenal index for sonographic quantification of liver steatosis. AJR Am J Roentgenol. 2009 Apr;192(4):909-14. doi: 10.2214/AJR.07.4016. PMID 19304694
- [Result] Labyed Y, Milkowski A. Novel Method for Ultrasound-Derived Fat Fraction Using an Integrated Phantom. J Ultrasound Med. 2020 Dec;39(12):2427-2438. doi: 10.1002/jum.15364. Epub 2020 Jun 11. PMID 32525261
- [Result] Gao J, Wong C, Maar M, Park D. Reliability of performing ultrasound derived SWE and fat fraction in adult livers. Clin Imaging. 2021 Dec;80:424-429. doi: 10.1016/j.clinimag.2021.08.025. Epub 2021 Sep 17. PMID 34543866